CLINICAL TRIAL: NCT00660335
Title: Phase III Study to Demonstrate the Efficacy and Safety of RG1068 (Synthetic Human Secretin)- Enhanced Magnetic Resonance Cholangiopancreatography (MRCP) in the Evaluation of Subjects With a History of Acute or Acute Recurrent Pancreatitis
Brief Title: Safety and Efficacy of Synthetic Human Secretin-Enhanced MRCP in Subjects With Abnormalities of the Pancreas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repligen Corporation (Industry)
Responsible Party: Melinda Livingstone, Repligen Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RG1068-16
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Pancreatitis
Keywords: secretin, RG1068, MRCP, pancreas
MeSH Terms: conditions — Pancreatitis | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG1068 (synthetic human secretin)

INTERVENTIONS:
Drug: RG1068 (synthetic human secretin) — Single-dose, IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of RG1068 (synthetic human secretin) with MRCP in subjects with abnormalities of the pancreas.

ELIGIBILITY:
Inclusion Criteria:

* History of pancreatitis
* Medically stable
* Able to give informed consent

Exclusion Criteria:

* Prior history of pancreatic resection
* Prior history of pancreatic duct drainage procedure
* Presence of a pancreatic stent
* Unstable cardiovascular disease
* Any contraindication to MRI procedure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-03; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be assessed by comparing baseline MRCP images and RG1068-enhanced MRCP images for the presence or absence of pancreatic abnormalities. | 0 - 10 minutes post dose

SECONDARY OUTCOMES:
The secondary outcome measure will assess safety | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David R Jacoby, MD, PhD, Study Director — Repligen Corporation

REFERENCES:
- [Derived] Sherman S, Freeman ML, Tarnasky PR, Wilcox CM, Kulkarni A, Aisen AM, Jacoby D, Kozarek RA. Administration of secretin (RG1068) increases the sensitivity of detection of duct abnormalities by magnetic resonance cholangiopancreatography in patients with pancreatitis. Gastroenterology. 2014 Sep;147(3):646-654.e2. doi: 10.1053/j.gastro.2014.05.035. Epub 2014 Jun 4. PMID 24906040